CLINICAL TRIAL: NCT06423586
Title: Positive Effect of Lecithin-based Delivery Form of Curcuma and Boswellia Extracts on Post-acute COVID-19 Irritable Bowel Syndrome. Two Cohorts of an Open-label Study.
Brief Title: Effect of Lecithin-based Curcuma and Boswellia on Post-acute COVID-19 IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0912/09052020
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Post-Acute COVID-19 Syndrome; Irritable Bowel Syndrome; Abdominal Pain; Dysbiosis
Keywords: abdominal pain; Bloating; Boswellia serrata; Covid-19 infection; Curcuma longa; Dysbiosis; IBS (irritable bowel syndrome); Long Covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Irritable Bowel Syndrome; Abdominal Pain; Dysbiosis; COVID-19 | interventions — turmeric extract

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCIBS Group (Experimental): Participants with post-acute COVID-19 irritable bowel syndrome (PCIBS) supplemented with lecithin-based formulations of Curcuma longa (Meriva™) and Boswellia serrata (Casperome™) extracts.
  Interventions: Dietary Supplement: Curcuma longa and Boswellia serrata extracts
- IBS Control Group (Active Comparator): Participants with irritable bowel syndrome (IBS) without prior COVID-19 infection supplemented with lecithin-based formulations of Curcuma longa (Meriva™) and Boswellia serrata (Casperome™) extracts.
  Interventions: Dietary Supplement: Curcuma longa and Boswellia serrata extracts

INTERVENTIONS:
Dietary Supplement: Curcuma longa and Boswellia serrata extracts — Participants received 500 mg of Curcuma longa and 150 mg of Boswellia serrata extracts (Meriva™ and Casperome™) twice daily for 30 days.

SUMMARY:
This open-label study investigates the effects of lecithin-based formulations of Curcuma longa (Meriva™) and Boswellia serrata (Casperome™) extracts on post-acute COVID-19 irritable bowel syndrome (PCIBS) and irritable bowel syndrome (IBS) without prior COVID-19 infection. A total of 44 participants, 16 with PCIBS and 28 controls with IBS, were supplemented for 30 days. Outcomes measured included abdominal bloating, abdominal pain, enteral dysbiosis, and global assessment of efficacy. The study found significant reductions in bloating and pain in both groups, with a notable decrease in dysbiosis only in the IBS group. This suggests potential benefits of the supplementation in managing gastrointestinal symptoms associated with PCIBS and IBS.

DETAILED DESCRIPTION:
This study aims to evaluate the efficacy and safety of lecithin-based formulations of Curcuma longa (Meriva™) and Boswellia serrata (Casperome™) extracts in treating gastrointestinal symptoms in patients with post-acute COVID-19 irritable bowel syndrome (PCIBS) and irritable bowel syndrome (IBS) without prior COVID-19 infection. The study was conducted at the Department of Public Health of the University of Pavia, Italy. Participants included 16 PCIBS patients and 28 IBS controls, aged 18-75 years. They were administered 500 mg of Curcuma longa and 150 mg of Boswellia serrata extracts twice daily for 30 days, in conjunction with a low FODMAP diet. Key outcomes measured were reductions in abdominal bloating and pain, changes in enteral dysbiosis as indicated by urinary indican levels, and overall treatment efficacy as assessed by participants. The study found that both groups experienced significant reductions in abdominal bloating and pain. However, a notable decrease in enteral dysbiosis was observed only in the IBS control group. The treatment was well tolerated with no reported adverse effects. These findings suggest that the combination of Curcuma longa and Boswellia serrata extracts may provide significant benefits in managing gastrointestinal symptoms associated with PCIBS and IBS.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years, male or female.
* Diagnosis of post-acute COVID-19 irritable bowel syndrome (PCIBS) 60-120 days after the end of infection.
* Diagnosis of irritable bowel syndrome (IBS) without prior COVID-19 infection.
* Evidence of functional abdominal bloating/distention (FAB/D) type of IBS according to Mearin et al.
* Presence of enteral dysbiosis defined by increased urinary indican values with normal skatole urinary concentration.

Exclusion Criteria:

* Normal urinary indican values or increased urinary skatole values.
* Subjects already on a low FODMAP diet or other dietary restrictions such as gluten-free diet or lactose-free diet within the past 6 months.
* Allergies to soy, nuts, or seafood, or insulin-dependent diabetes.
* Known history of celiac disease, symptomatic diverticular disease, inflammatory bowel disease, or microscopic colitis.
* Prior small bowel or colonic surgery or cholecystectomy.
* Presence of bloody diarrhea or severe vomiting.
* Severe renal disease (serum creatinine >1.5 mg/dL) or liver disease (altered liver function tests).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Reduction in Abdominal Bloating | 30 days
  Measure the change in abdominal bloating severity from baseline to the end of the study using a validated questionnaire.

SECONDARY OUTCOMES:
Change in Urinary Indican Levels | 30 days
  Evaluate the change in urinary indican levels from baseline to the end of the study to assess enteral dysbiosis

OTHER OUTCOMES:
Global Assessment of Efficacy (GAE) | 30 days
  Assess the overall efficacy of the treatment using a 4-point scale (ineffective, moderately effective, effective, very effective).

CONTACTS AND LOCATIONS:
Overall Officials: Giacosa Attilio, Principal Investigator — Italian Diagnostic Center (CDI)
Locations (1):
- Mariangela Rondanelli, Pavia, PV, Italy

IPD SHARING:
Plan to Share IPD: No